CLINICAL TRIAL: NCT03676335
Title: A Phase Ⅱ, Multicenter, Randomized, Single-blind, Positive-controlled, Dose-finding Study to Assess the Efficacy and Safety of CsA Ophthalmic Gel in Subjects With Moderate to Severe Aqueous-Deficient Dry Eye (ADDE)
Brief Title: Assess the Safety and Efficacy of CsA Ophthalmic Gel in Subjects With Dry Eye
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Zhaoke (Guangzhou) Ophthalmology Pharmaceutical Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ZK-CSA-201704
Record Dates: First submitted 2018-08-30; First posted 2018-09-18 (Actual); Last update posted 2020-05-08 (Actual); Status verified 2020-05

CONDITIONS: Dry Eye
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- 0.3 g: 0.15 mg（1)&Hypromellose Eye Drops (Experimental): Sixty subjects will be treated with CsA eye gel: 0.3 g: 0.15 mg, 1 times daily, The treatment period is 12 weeks. The basic medicine is Hypromellose Eye Drops, 3 times daily for 12 weeks.
  Interventions: Drug: CsA eye gel; Drug: Hypromellose Eye Drops
- 0.3 g: 0.15mg（2)&Hypromellose Eye Drops (Experimental): Sixty subjects will be treated with CsA eye gel: 0.3 g: 0.15 mg, 2 times daily, interval of about 12 hours, The treatment period is 12 weeks. The basic medicine is Hypromellose Eye Drops, 3 times daily for 12 weeks.
  Interventions: Drug: CsA eye gel; Drug: Hypromellose Eye Drops
- 0.3 g: 0.3 mg &Hypromellose Eye Drops (Experimental): Sixty subjects will be treated with CsA eye gel: 0.3 g: 0.3 mg, 1 times daily, The treatment period is 12 weeks. The basic medicine is Hypromellose Eye Drops, 3 times daily for 12 weeks.
  Interventions: Drug: CsA eye gel; Drug: Hypromellose Eye Drops
- 0.4 ml: 0.2 mg &Hypromellose Eye Drops (Active Comparator): Sixty subjects will be treated with CsA for eye emulsion: 0.4 ml: 0.2 mg, 2 times daily, interval of about 12 hours, The treatment period is 12 weeks. The basic medicine is Hypromellose Eye Drops, 3 times daily for 12 weeks.
  Interventions: Drug: CsA for eye emulsion; Drug: Hypromellose Eye Drops

INTERVENTIONS:
Drug: CsA eye gel — The CsA eye gel of 0.3 g: 0.15 mg, 0.3 g: 0.3 mg
  Other Names: CsA gel
  Arms: 0.3 g: 0.15 mg（1)&Hypromellose Eye Drops; 0.3 g: 0.15mg（2)&Hypromellose Eye Drops; 0.3 g: 0.3 mg &Hypromellose Eye Drops
Drug: CsA for eye emulsion — The CsA for eye emulsion of 0.4 ml: 0.2 mg
  Other Names: CsA emulsion
  Arms: 0.4 ml: 0.2 mg &Hypromellose Eye Drops
Drug: Hypromellose Eye Drops — Hypromellose Eye Drops of 15ml：75mg, 3 times daily, 1-2 drop
  Other Names: zhenshishuang

SUMMARY:
The purpose of this study is to explore the efficacy and safety of CsA ophthalmic gel in the treatment of moderate to severe tear deficiency dry eye with different dosage, frequency and concentration, and to preliminarily determine the optimal dosage, frequency and concentration, so as to provide a theoretical basis for the design of follow-up clinical studies.

DETAILED DESCRIPTION:
A multicenter, randomized, single-blind, positive controlled exploratory study will be conducted with cyclosporine A ophthalmic emulsion as the control drug.

The experimental drugs were divided into three groups:

Treatment group A: CsA eye gel: 0.3 g: 0.15 mg, once daily； Treatment group B: CsA eye gel: 0.3 g: 0.15 mg, twice daily, interval of about 12 hours； Treatment group C: CsA eye gel: 0.3 g: 0.3 mg, once daily. One drop into each eye when you use it.

Control group: CsA emulsion: 0.4 ml: 0.2 mg. One drop into the eye, 2 times daily with an interval for 12 hours.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18, both male and female;
2. Pregnancy tests were negative for women of childbearing age and contraceptive measures (including abstinence, intrauterine devices, diaphragms and spermicides) were taken during the trial. Men are willing to use approved contraceptive methods (possibly using condoms and spermicides or oral contraceptives, implants or injections of contraceptives, intrauterine devices, diaphragms and spermicides) or sexual partner infertility;
3. According to the symptoms and signs and ophthalmologic examinations, the patients were diagnosed as moderate to severe dry eye;

   1. EDS score is more than 40 points;
   2. BUT is less than 10 s;
   3. Schirmer test result is less than 10mm/5 min;
   4. In any area, corneal fluorescein staining was more than 2 points.
4. The anatomy of the eyelids is normal and has normal blinking function;
5. Patients with newly diagnosed dry eye disease, or who are undergoing dry eye treatment, voluntarily discontinue treatment within 72 hours of entering the screening period;
6. Ability and willingness to participate in all research assessments and all planned visits during the pilot period in accordance with the programme requirements;
7. Agree to participate in the study and voluntarily sign informed consent.

Exclusion Criteria:

1. Allergy to CsA, fluorescein or any component of the drug is known;
2. Severe dry eye patients requiring surgical treatment;
3. Glaucoma patients;
4. Unwilling to avoid wearing contact lenses;
5. Within 12 months prior to the start of the study, intraocular surgery or internal surgery was necessary;
6. Eyelid surgery was performed within 6 months prior to the start of the study, or dry eye secondary to surgery;
7. Those who had undergone corneal refractive surgery or keratoplasty;
8. Congenital lacrimal gland or meibomian gland deficiency or lacrimal gland obstructive diseases;
9. Systemic inflammation or active eye infection and blepharitis;
10. Patients with ocular cicatricial pemphigoid, obvious conjunctival scar, ocular chemical burn and neurotrophic keratoconjunctivitis;
11. Who suffered from ocular malignancies;
12. No other eye drops could be stopped during the study period;
13. Systemic or uncontrollable disorders that affect the collection of research parameters or patient compliance, such as severe cardiopulmonary disease, uncontrollable hypertension and diabetes;
14. With history of central nervous system disease or epilepsy, and / or mental disorder;
15. Pregnant women and lactating women, or women of childbearing age, do not adopt effective contraceptive measures;
16. Participated in other clinical trials or participated in other clinical trials within 1 months before the election;
17. Systemic or topical cyclosporine drugs within 3 months;
18. Patients who were not considered suitable for the study, including those who were unable or unwilling to comply with the protocol requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2018-05-09 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-12-12 (Actual)

PRIMARY OUTCOMES:
The EDS score at the NO.5 visit was compared with the baseline EDS score (binocular) | 84 days after admission
  0-100 points VAS score was evaluated

SECONDARY OUTCOMES:
The EDS score at the NO.3, NO.4 visit were compared with the baseline EDS score (binocular) | 14 days after admission ，42days after admission
  0-100 points VAS score was evaluated
Average changes in VAS scores of 6 dry eye symptoms (burning/needling sensation, pruritus, foreign body sensation, discomfort, photophobia and pain) at the NO.3, NO.4 and NO.5 visit were compared with baseline (binocular) | 14 days after admission ，42 days after admission ，84days days after admission
  0-100 points VAS score was evaluated
Comparison of the NO.3, NO.4, NO.5 visit and baseline corneal fluorescein staining changes | 14 days after admission ，42 days after admission ，84 days after admission
  score（The cornea was divided into five quadrants: central, upper, lower, temporal and nasal. The cornea was stained with 4 points, 0 points for non-staining, 1 point for scattered dotted staining, 2 points for clan staining, 3 points for local dense + scattered dotted staining and 4 points for extensive diffuse staining. The total score is the sum of the quadrant scores）
Comparison of the NO.3, NO.4, NO.5 visit and baseline BUT changes | 14 days after admission ，42 days after admission ，84 days after admission
  time
Comparison of the NO.3, NO.4, NO.5 visit and baseline Schirmer changes | 14 days after admission ，42 days after admission ，84 days after admission
  Basal tear secretion

CONTACTS AND LOCATIONS:
Overall Officials: shiyou zhou, PHD, Study Director — Ophthalmological Center of Zhongshan University
Locations (1):
- Ophthalmological Center of Zhongshan University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Utine CA, Stern M, Akpek EK. Clinical review: topical ophthalmic use of cyclosporin A. Ocul Immunol Inflamm. 2010 Oct;18(5):352-61. doi: 10.3109/09273948.2010.498657. PMID 20735287
- [Result] Kunert KS, Tisdale AS, Gipson IK. Goblet cell numbers and epithelial proliferation in the conjunctiva of patients with dry eye syndrome treated with cyclosporine. Arch Ophthalmol. 2002 Mar;120(3):330-7. doi: 10.1001/archopht.120.3.330. PMID 11879137
- [Result] Kim EC, Choi JS, Joo CK. A comparison of vitamin a and cyclosporine a 0.05% eye drops for treatment of dry eye syndrome. Am J Ophthalmol. 2009 Feb;147(2):206-213.e3. doi: 10.1016/j.ajo.2008.08.015. Epub 2008 Oct 9. PMID 18848318
- [Result] Barr JT, Schechtman KB, Fink BA, Pierce GE, Pensyl CD, Zadnik K, Gordon MO. Corneal scarring in the Collaborative Longitudinal Evaluation of Keratoconus (CLEK) Study: baseline prevalence and repeatability of detection. Cornea. 1999 Jan;18(1):34-46. PMID 9894935
- [Result] Research in dry eye: report of the Research Subcommittee of the International Dry Eye WorkShop (2007). Ocul Surf. 2007 Apr;5(2):179-93. doi: 10.1016/s1542-0124(12)70086-1. PMID 17508121